CLINICAL TRIAL: NCT07053228
Title: e-Natureza Blue Care - Impact of Virtual Reality on Pain Perception, Mood States, and Analgesic Use in Patients With Cancer Pain: Randomized Clinical Trial.
Brief Title: e-Natureza Blue Care: Nature-based Virtual Reality and Pain Perception
Acronym: e-NatBlue
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Eliseth Ribeiro Leao, Nurse Scientist, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 86844425.5.0000.0071
Record Dates: First submitted 2025-06-24; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Cancer Pain; Palliative Care
Keywords: Cancer Pain; Palliative care; Virtual reality
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial, an experimental study involving human subjects aimed at evaluating the effect of a health-related intervention. After signing the informed consent form, participants will be randomly assigned via the Randomizer software to either the control or intervention group. Patients in the control group will receive standard pain management, which includes pharmacological treatment and monitoring through electronic medical records (EMRs). When pain is not adequately controlled, the institutional Pain Management Team conducts an in-depth EMR review to tailor care, ensuring effective and continuous pain relief. The intervention group will receive standard care plus immersive nature-based virtual reality therapy. Five tools will be used for data collection: a Sociodemographic and Clinical Questionnaire, the Visual Analogue Scale , the Positive and Negative Affect Schedule , the Nature Connectedness Scale (NCS), and the Analgesic Experience Questionnaire
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Nature-based Virtual Reality (Experimental): Participants will view an 8-minute 360° 3D immersive video featuring natural Brazilian blue environments (beach, waterfall) developed using the Oculus Go. Pre- and post-intervention assessments will include: Visual Analog Scale (VAS), The Positive and Negative Affect Schedule (PANAS), After 24h, the Analgesic Experience Form will be completed. A sociodemographic/clinical questionnaire and Connectedness to Nature Scale (CNS) will be applied only pre-intervention.
  Interventions: Behavioral: Nature-based virtual reality
- Control (Active Comparator): Participants in the control group will receive standard care. They will undergo standard pain management as per institutional pain protocols. The same outcomes assessment will occur at the same time intervals as in the intervention group.
  Interventions: Drug: Standard Pain Management

INTERVENTIONS:
Behavioral: Nature-based virtual reality — Participants in this group will receive standard pain management care plus one session of immersive virtual reality (VR) using Oculus Go headsets. The session consists of viewing a nature-themed 360º video (e.g., beach, waterfall, songbirds) for approximately 8 minutes, accompanied by synchronized natural sounds.
  The VR experience is designed to promote distraction, relaxation, and emotional engagement with nature to support pain relief and emotional regulation. The equipment is sanitized between uses according to hospital infection control protocols.
  Other Names: Non-pharmacological pain relief
  Arms: Intervention - Nature-based Virtual Reality
Drug: Standard Pain Management — Participants in this group will receive the institution's standard pharmacological pain management, monitored and adjusted by the Pain Control Team using the hospital's electronic medical record system. This may include opioid and non-opioid analgesics according to clinical evaluation.
  No complementary interventions will be provided during the study period.
  Other Names: Pharmacological pain relief
  Arms: Control

SUMMARY:
This randomized clinical trial aims to evaluate the effectiveness of immersive nature-based virtual reality in managing chronic pain among oncology patients. The study seeks to expand non-pharmacological treatment options and contribute to the therapeutic arsenal available for chronic pain management in cancer care.The intervention utilizes immersive videos of diverse Brazilian natural environments to promote analgesic and emotional relief.

DETAILED DESCRIPTION:
Pain is a global health issue and remains the most feared symptom among cancer patients. With over 14 million new cancer diagnoses annually and projections suggesting this number will triple by 2030. The majority of patients are diagnosed at an advanced stage, where pain is the predominant complaint. The concept of total pain, as described in palliative care, highlights the need for a multidimensional approach that addresses physical, psychological, social, and spiritual aspects.

In the management of chronic pain, complementary therapies such as acupuncture, meditation, and massage have gained prominence for offering holistic benefits without the side effects associated with pharmacological treatments. Another promising complementary approach involves exposure to natural environments. Immersive Virtual Reality (VR) is an innovative strategy that provides distraction and reduces pain perception by transporting patients to engaging, nature-based virtual settings.

This study is a randomized, controlled, parallel-group clinical trial designed to investigate the impact of an immersive virtual reality (VR) intervention with nature-themed content (blue spaces) on pain and emotional well-being in hospitalized cancer patients. The research will be conducted in three oncology units of a large private hospital in São Paulo, Brazil.

A total of 130 adult oncology inpatients experiencing chronic pain will be randomly assigned to either the intervention or control group. Participants in the control group will receive standard pain management as provided by the hospital's pain control team, guided by electronic medical records, and institutional pain protocols. The intervention group will receive the same standard care, plus a VR session using the Oculus Go headset and 360-degree nature videos with synchronized natural sounds (e.g., beach, waterfall, birdsong), lasting approximately 8 minutes.

Data will be collected using the following validated instruments:

Visual Analog Scale (VAS) for pain intensity,

PANAS for positive and negative affect,

Nature Connectedness Scale (NCS),

Sociodemographic and clinical questionnaire,

Analgesic Use Form, developed by researchers to quantify medication use and pharmacological class.

Ethical approval was obtained (CAAE: 86844425.5.0000.0071), and all participants will provide written informed consent. If the results are positive, the intervention will be made available to the hospital's pain management team for broader implementation in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized oncological patients with chronic pain.
* both sexes
* aged 18 years or older
* preserved clinical condition and communication abilities that allow participation in the study
* report pain documented in the electronic medical record

Exclusion Criteria:

* Patients who are unable to tolerate wearing the virtual reality (VR) headset for at least 8 minutes
* blind patients
* patients who experience any side effects or worsening clinical condition during the interview/intervention period
* patients undergoing other complementary treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogic Scale for Pain | Immediately post-intervention for an unique virtual reality intervention
  Change from Baseline in self-reported pain intensity using a 0-10 Visual Analog Scale at post intervention. Will be applied the Visual Analogue Scale - VAS. It is one of the most used instruments for pain assessment with a score from 0 to 10 that allows the patient to evaluate the pain of the procedure through a visual analogue scale numbered from zero to ten, with zero no pain, ten being the worst pain ever felt in life.
Frequency of analgesic administration Frequency of analgesic administration Frequency of analgesic administration | 24 hours post-intervention
  This outcome will assess the number of doses of analgesics administered to participants in the control and experimental groups within 24 hours following each intervention session. Analgesics include opioids, non-opioids, and adjuvant medications. Data will be collected from medical records.
Total dosage of analgesics administered | 24 hours post-intervention
  This outcome will assess and compare the total dosage (in milligrams) of analgesics administered to participants in the control and experimental groups within 24 hours after each intervention session. The analysis will include opioids, non-opioids, and adjuvant medications. Data will be extracted from medical records.
Type of analgesics administered | 24 hours post-intervention
  This outcome will identify and compare the types of analgesics (opioids, non-opioids, and adjuvant medications) used by participants in the control and experimental groups within 24 hours following each intervention session. Medication classes will be categorized based on pharmacological criteria.

SECONDARY OUTCOMES:
The Positive and Negative Affect Schedule (PANAS) | Immediately post-intervention for an unique virtual reality intervention
  Change from Baseline Affective States at post-intervention. PANAS is a 20-item self- report measure to assess positive affect (PA) and negative affect (NA). It is one of the most used instruments in the investigation of affective states composed of 20 questions and each item can be rated on a likert type frequency scale of sensations, ranging from 0 (not at all) to 5 (extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Eliseth R Leão, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelleher SA, Fisher HM, Winger JG, Miller SN, Amaden GH, Somers TJ, Colloca L, Uronis HE, Keefe FJ. Virtual reality for improving pain and pain-related symptoms in patients with advanced stage colorectal cancer: A pilot trial to test feasibility and acceptability. Palliat Support Care. 2022 Aug;20(4):471-481. doi: 10.1017/S1478951521002017. PMID 35078545
- [Background] Britton E, Kindermann G, Domegan C, Carlin C. Blue care: a systematic review of blue space interventions for health and wellbeing. Health Promot Int. 2020 Feb 1;35(1):50-69. doi: 10.1093/heapro/day103. PMID 30561661

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-04-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT07053228/Prot_ICF_000.pdf